CLINICAL TRIAL: NCT04973735
Title: A Phase I, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of LY-CovMab Injection in Chinese Healthy Subjects
Brief Title: A Phase I Study of LY-CovMab Injection in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY-CovMab/CT-CHN-101
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 30mg LY-CovMab (Experimental): LY-CovMab is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab
- 150mg LY-CovMab (Experimental): LY-CovMab is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab
- 600mg LY-CovMab (Experimental): LY-CovMab is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab
- 1200mg LY-CovMab (Experimental): LY-CovMab is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab
- 2400mg LY-CovMab (Experimental): LY-CovMab is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab
- Placebo (Placebo Comparator): Placebo is diluted with 0.9% sodium chloride to a total volume of 250 mL for IV infusion
  Interventions: Drug: LY-CovMab

INTERVENTIONS:
Drug: LY-CovMab — single IV infusion

SUMMARY:
A single center, randomized, doubled-blind, placebo-control and single ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of LY-CovMab Injection in Chinese healthy subjects.

DETAILED DESCRIPTION:
A single center, randomized, doubled-blind, placebo-control and single ascending dose phase I study:

Primary objective: to evaluate the safety and tolerability of a single dose of LY-CovMab Injection in Chinese healthy subjects.

Secondary objective: to evaluate the pharmacokinetics (PK) and immunogenicity of a single dose of LY-CovMab injection in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

A signed informed consent form (ICF) from the patient or their legally authorized representative.

Healthy males or females, ages ≥18 to ≤45 years. Male subjects with weight ≥50 kg, or female subjects with weight ≥45 kg, and body mass index (BMI) 19.0≤BMI≤26.0 kg/m2.

No abnormality, or no clinically significant abnormality in vital signs, physical examination, laboratory tests, and 12-lead ECG in Chinese healthy subjects during the screening period.

Female patients of childbearing potential (defined as female subjects who do not receive any operative sterilization or who had been through menopause for less than 1 year) must have a negative result for pregnancy test at screening. Male and female subjects with childbearing potential must agree to adopt effective contraceptive methods at least from 2 weeks prior to screening to 6 months after administration of the investigational drug.

Exclusion Criteria:

Those who have had surgery within 8 weeks prior to screening or who have surgery planned during the trial, and the investigator believes that such surgery may bring potential risks to the subjects.

Prior to administration of the investigational drug, use of the following drugs or therapies:

i. any prescription drug within 28 days. ii. any over-the-counter drug, including health care products within 7 days.

Prior history or current evidence of serious disease or chronic disease of the respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, immune system, hematology, psychiatry, and dermatology, etc, or any disease that may interfere with the trial results.

Subjects with coronavirus disease 2019 (COVID-19) or recovered from it or subjects positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleic acid or serum SARS-CoV-2 specific antibodies.

Subjects who are with known history of allergies to any ingredient of the investigational drug, or similar drugs, or subjects with allergic constitution (previously sensitive to ≥ 2 foods or drugs).

Subjects with any positive test of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, treponema pallidum antibody, or human immunodeficiency virus (HIV) antibody.

Subjects with alcohol abuse or tobacco abuse, or alcohol blood test results exceeding the upper limit of the normal range. Alcohol abuse is defined as: alcohol consumption of more than 14 U (1 U = 350 mL of beer, or 45 mL of liquor, or 150 mL of wine) per week within 3 months prior to screening. Tobacco abuse is defined as: smoking ≥5 cigarettes per day on average within 3 months prior to screening.

Female subjects (including partners) who plan to be pregnant within one year upon screening, or pregnant or breast-feeding female subjects.

Subjects with a history of drug addiction or drug abuse, or with positive urine screen test results for drug.

Subjects donating whole blood or blood components, or with massive hemorrhage (>400 mL), within 3 months prior to screening.

Prior vaccination with SARS-CoV-2 vaccine or participation in a SARS-CoV-2 neutralizing antibody clinical trial. Participation in any other clinical study with pharmacological intervention within 3 months prior to screening, or the drug is still within the elimination period (5 half-lives) prior to screening, whichever is longer. Vaccination within 12 weeks prior to screening, or planned vaccination during the study and within 12 weeks after the end of the study.

Subjects with a history of fainting at the sight of blood or puncture. Subjects who are not suitable to participate in the clinical trial as considered by the investigator or cannot complete the study for any other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Changes in Body Temperature | up to 99 days
  Grade of treatment-emergent changes in body temperature by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent Changes in Respiratory Rate | up to 99 days
  Grade of treatment-emergent changes in respiratory rate by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent Changes in Pulse Rate | up to 99 days
  Grade of treatment-emergent changes in pulse rate by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent Changes in Blood Pressure | up to 99 days
  Grade of treatment-emergent changes in blood pressure by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Safety Laboratory Value (Haematology) | D-1, D4, D8, D15, D29, D50, D99
  Haematology laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Safety Laboratory Value (blood chemistry) | D-1, D4, D8, D15, D29, D50, D99
  Serum Chemistry laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Frequency and Grade of Adverse Events | up to 99 days
Assess safety profile of LY-CovMab | D-1, D4, D8, D15, D29, D50, D99
  12 lead electrocardiogram (ECG) heart rate
Assess safety profile of LY-CovMab | D-1, D4, D8, D15, D29, D50, D99
  12 lead electrocardiogram (ECG) PR interval
Assess safety profile of LY-CovMab | D-1, D4, D8, D15, D29, D50, D99
  12 lead electrocardiogram (ECG) QTc interval
Assess safety profile of LY-CovMab | D-1, D4, D8, D15, D29, D50, D99
  12 lead electrocardiogram (ECG) QRS interval

SECONDARY OUTCOMES:
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Maximum observed concentration (Cmax)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Time to maximum observed concentration (Tmax)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0 last)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Percentage of the extrapolated area under the concentration-time curve (AUC_%Extrap)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Area under the concentration-time curve from time 0 to infinity (AUC0-inf),
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Clearance (CL)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Half-life (t1/2)
Assess Pharmacokinetic parameters of LY-CovMab | up to 99 days
  Volume of distribution (Vd)
Assess the immunogenicity of LY-CovMab | D1, D15, D29, D43, D57, D71, D99
  Incidence of anti-drug antibody (ADA)
Assess the immunogenicity of LY-CovMab | D1, D15, D29, D43, D57, D71, D99
  Incidence of neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, Dr, Principal Investigator — The Second Hospital of Anhui Medical University; Wei Hu, Dr, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Zhou R, Yang J, Dou C, Gan T, Liu F, Hu B, Song D, Lu C, Hu W. A Randomized, Double-Blind, Placebo-Controlled, First-in-Human Clinical Trial to Assess Safety, Tolerability, and Pharmacokinetics of LY-CovMab, a Potent Human Neutralizing Antibody Against SARS-CoV-2. Infect Dis Ther. 2022 Feb;11(1):405-422. doi: 10.1007/s40121-021-00572-x. Epub 2021 Dec 8. PMID 34878625